CLINICAL TRIAL: NCT02990728
Title: Mirena® ± Metformin as Fertility-preserving Treatment for Young Asian Women With Early Endometrial Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ting-Chang Chang, Director, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTC-184
Record Dates: First submitted 2016-11-16; First posted 2016-12-13 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Endometrial Cancer
Keywords: Endometrial Cancer.Mirena®
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mirena® + metformin (Experimental): The enrolled patient is allocated to either LNG-IUS only or LNG-IUS + metformin by central randomization with study site allocation. A 90-100 days of continuous treatment before first histologic assessment of treatment response is required. The patient will receive endometrial curettage or hysteroscopic evaluation and resection of suspected lesion after 90-100 days of treatment. Patients with good response to assigned treatment will continue the treatment for another 90-100 days and second histologic assessment will be performed. Patients with poor response to assigned treatment at first assessment will receive additive oral progestin therapy, along with the assigned regimen(s) as, Oral progestin, either medroxyprogesterone acetate 500 mg daily or oral megestrol acetate 160 mg daily After a total of at least 6 months treatment period, the patient with good response at first assessment is suggested to keep the Mirena for maintenance until plan to get pregnant
  Interventions: Drug: Metformin; Device: Mirena®
- Mirena® (Active Comparator): The enrolled patient is allocated to either LNG-IUS only or LNG-IUS + metformin by central randomization with study site allocation. A 90-100 days of continuous treatment before first histologic assessment of treatment response is required. The patient will receive endometrial curettage or hysteroscopic evaluation and resection of suspected lesion after 90-100 days of treatment. Patients with good response to assigned treatment will continue the treatment for another 90-100 days and second histologic assessment will be performed. Patients with poor response to assigned treatment at first assessment will receive additive oral progestin therapy, along with the assigned regimen(s) as, Oral progestin, either medroxyprogesterone acetate 500 mg daily or oral megestrol acetate 160 mg daily After a total of at least 6 months treatment period, the patient with good response at first assessment is suggested to keep the Mirena for maintenance until plan to get pregnant
  Interventions: Device: Mirena®

INTERVENTIONS:
Drug: Metformin — The enrolled patient is allocated to either LNG-IUS only or LNG-IUS + metformin by central randomization with study site allocation. A 90-100 days of continuous treatment before first histologic assessment of treatment response is required. The patient will receive endometrial curettage or hysteroscopic evaluation and resection of suspected lesion after 90-100 days of treatment. Patients with good response to assigned treatment will continue the treatment for another 90-100 days and second histologic assessment will be performed. Patients with poor response to assigned treatment at first assessment will receive additive oral progestin therapy, along with the assigned regimen(s) as, Oral progestin, either medroxyprogesterone acetate 500 mg daily or oral megestrol acetate 160 mg daily After a total of at least 6 months treatment period, the patient with good response at first assessment is suggested to keep the Mirena for maintenance until plan to get pregnant
  Arms: Mirena® + metformin
Device: Mirena®

SUMMARY:
Primary objective To discover the efficacies of levonorgestrel-containing intrauterine device (LNG-IUS, Mirena®), with or without metformin, as fertility-preserving treatment for grade 1 endometrioid adenocarcinoma of endometrium, cT1aN0M0 with presumed no myometrial invasion on image study (MRI preferred).

Secondary objectives

1. To discover the morphological and molecular change in the endometrium tumor before and after treatment
2. To discover the effectiveness of adding oral progestin to subjects who show no good response to assigned
3. To compare (1) the systemic effects, including body weight change, neuropsychiatric alternation, GI disturbance, skin disorder, change in serum metabolic and hepatic markers between the two study patient groups; (2) The rate of long-term success defined as (a) sustained remission of >= 12 months starts from the histologic documentation of complete remission (b) rate of pregnancy and (c) alive baby delivery, based on time-to-event analysis.
4. Molecular markers and their expression before, during and after treatment, including progesterone B receptor, progesterone A receptor, estrogen receptor, Ki67, PTEN and its related markers, Bcl2 and its related markers and other developing markers. This is to discover prediction markers to medical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Women <= 40 years old with histologic confirmed grade 1 endometrioid adenocarcinoma of the endometrium
2. Tumour is confirmed to the endometrial cavity with no evidence of metastasis on MRI and/or trans-vaginal ultrasonography
3. ECOG 0-1, adequate organ function, with fertility preserving need
4. Immunohistochemical study showed positive progesterone receptor and positive estrogen receptor in the endometrial tumour tissue
5. Serum CA 125 titre is within normal limit
6. Signed informed consent

Exclusion Criteria:

1. Women age > 40 years or endometrial cancer other than grade 1 endometrioid adenocarcinoma
2. Suspected lymph node metastasis or other metastasis appears in image study
3. Ovarian tumour in image study
4. Blurred junction between the endometrium and the myometrium on image study, with the impression that myometrial invasion of the endometrial tumour cannot be ruled out
5. Ultrasonographic study or MRI show obvious adenomyosis or ovarian endometriosis
6. Women who are contraindicated to receive study treatment because of intolerance to treatment agents, medical co-morbidity or other reason(s)
7. Women with history of or concurrent with malignancy other than skin basal cell carcinoma
8. Women who cannot participate regular follow-up

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2016-03; Primary Completion 2018-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
the efficacies of levonorgestrel-containing intrauterine device (LNG-IUS, Mirena®), with or without metformin | the efficacies of levonorgestrel-containing intrauterine device (LNG-IUS, Mirena®), with or without metformin about 6 month

IPD SHARING:
Plan to Share IPD: No